CLINICAL TRIAL: NCT03723096
Title: Expanded Access for CC-4047
Status: No longer available | Type: Expanded Access
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-4047
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Multiple Myeloma
Keywords: Expanded Access; Compassionate Use
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: CC-4047 — CC-4047 will be administered orally
  Other Names: Pomalyst, Pomalidomide

SUMMARY:
This is an expanded access program (EAP) for eligible participants designed to provide access to CC-4047.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Celgene, Summit, New Jersey, United States